CLINICAL TRIAL: NCT00264797
Title: Randomized Controlled Trial of Osmotic-Release Methylphenidate (OROS-MPH) for Attention Deficit Hyperactivity Disorder (ADHD) in Adolescents With Substance Use Disorders (SUD)
Brief Title: Attention Deficit Hyperactivity Disorder (ADHD) in Adolescents With Substance Use Disorders (SUD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Theresa Winhusen, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-CTN-0028; 5U10DA013732 (NIH)
Record Dates: First submitted 2005-12-10; First posted 2005-12-13 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-05

CONDITIONS: ADHD; Substance Abuse
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Active Comparator)
  Interventions: Drug: Methylphenidate (OROS-MPH)
- Methylphenidate (Placebo) (Placebo Comparator)
  Interventions: Drug: Methylphenidate (OROS-MPH) - Placebo

INTERVENTIONS:
Drug: Methylphenidate (OROS-MPH) — Participants will be scheduled for weekly medication (OROS-MPH) and research assessment visits (approximately 45 minutes to 1 hour in length). A forced titration dosing strategy will be used starting with 18 mg/day OROS-MPH for 3 days, increasing to 36mg/day for the next three days; increasing to 54 mg/day in week two, and to 72 mg/day in week three through the remainder of the study (as tolerated). Participants will also attend weekly CBT sessions (approximately 1 hour in length) targeting their drug use.
  Arms: Methylphenidate
Drug: Methylphenidate (OROS-MPH) - Placebo — Participants will be scheduled for weekly medication and research assessment visits (approximately 45 minutes to 1 hour in length). A forced titration dosing strategy will be used starting with 18 mg/day OROS-MPH placebo for 3 days, increasing to 36mg/day for the next three days; increasing to 54 mg/day in week two, and to 72 mg/day in week three through the remainder of the study (as tolerated). Participants will also attend weekly CBT sessions (approximately 1 hour in length) targeting their drug use.
  Arms: Methylphenidate (Placebo)

SUMMARY:
The purpose of this study is to determine the efficacy of osmotic-release methylphenidate (OROS-MPH) versus placebo for the treatment of ADHD in adolescents with SUD.

DETAILED DESCRIPTION:
Research shows a high prevalence of Attention Deficit Hyperactivity Disorder (ADHD) in adolescents with substance abuse disorders and indicates that they have poorer substance use treatment outcomes and poorer prognosis and risk of persistence and progression of drug use and behavior problems into adulthood. Although research indicates that the majority are not treated for ADHD while in substance treatment, we do not know whether concurrent pharmacotherapy for ADHD will improve treatment outcomes. This Clinical Trials Network (CTN) study will evaluate the efficacy of osmotic-release methylphenidate (OROS-MPH), relative to placebo, in treating ADHD and decreasing substance use in adolescents (13-18 years old) with ADHD and a substance use disorder. Approximately 300 participants will be recruited at 11 sites and randomly assigned to either OROS-MPH or matching placebo for a 16-week treatment period, during which all participants will receive individual cognitive-behavioral therapy as a standardized treatment for substance abuse.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual for Mental Disorders, 4th Edition (DSM-IV) diagnostic criteria for ADHD
* Meet DSM-IV diagnostic criteria for at least one non-nicotine substance use disorder
* Has a DSM-IV ADHD Symptom Checklist score ≥ 22 derived from the adolescent-completed checklist

Exclusion Criteria:

* Serious medical illness
* History of tic disorder
* Pregnant or breastfeeding
* Meet DSM-IV criteria for current or life-time psychotic disorder
* Meet DSM-IV criteria for current or life-time bipolar disorder
* Requires/or prescribed other concurrent psychotropic medication
* Taking any medications that may produce interactions with OROS-MPH
* Opiate dependence
* Methamphetamine abuse or dependence
* Suicidal risk
* Enrolled in an inpatient, residential, day treatment, or outpatient substance abuse program within 28 days prior to signing consent

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 303 (Actual)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Riggs, M.D., Principal Investigator — University of Colorado, Denver; Theresa Winhusen, Ph.D., Principal Investigator — University of Cincinnati
Locations (12):
- United States (12):
  - Synergy Treatment Center, Denver, Colorado
  - Gateway Community Services, Jacksonville, Florida
  - Operation PAR, Inc., St. Petersburg, Florida
  - Mountain Manor Treatment Programs, Baltimore, Maryland
  - SSTAR: Stanley Street Treatment & Resources, Inc, Fall River, Massachusetts
  - Crittenton, Kansas City, Missouri
  - St. Luke's-Roosevelt Hospital, Child and Family Institute, New York, New York
  - Rehab After Work-Life Counseling Services, Paoli, Pennsylvania
  - Addiction Medicine Services, Pittsburgh, Pennsylvania
  - SSTAR of Rhode Island, North Kingstown, Rhode Island
  - LRADAC, Columbia, South Carolina
  - Mental Health and Retardation of Tarrant County, Fort Worth, Texas

REFERENCES:
- [Background] Riggs PD, Winhusen T, Davies RD, Leimberger JD, Mikulich-Gilbertson S, Klein C, Macdonald M, Lohman M, Bailey GL, Haynes L, Jaffee WB, Haminton N, Hodgkins C, Whitmore E, Trello-Rishel K, Tamm L, Acosta MC, Royer-Malvestuto C, Subramaniam G, Fishman M, Holmes BW, Kaye ME, Vargo MA, Woody GE, Nunes EV, Liu D. Randomized controlled trial of osmotic-release methylphenidate with cognitive-behavioral therapy in adolescents with attention-deficit/hyperactivity disorder and substance use disorders. J Am Acad Child Adolesc Psychiatry. 2011 Sep;50(9):903-14. doi: 10.1016/j.jaac.2011.06.010. Epub 2011 Aug 4. PMID 21871372
- [Derived] Tamm L, Trello-Rishel K, Riggs P, Nakonezny PA, Acosta M, Bailey G, Winhusen T. Predictors of treatment response in adolescents with comorbid substance use disorder and attention-deficit/hyperactivity disorder. J Subst Abuse Treat. 2013 Feb;44(2):224-30. doi: 10.1016/j.jsat.2012.07.001. Epub 2012 Aug 11. PMID 22889694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted by the National Institute on Drug Abuse (NIDA) Clinical Trials Network (CTN) between March 2006 and October 2008. Eleven community based treatment programs recruited participants.
Groups:
- Methylphenidate: Methylphenidate (OROS-MPH) : Participants will be scheduled for weekly medication (OROS-MPH) and research assessment visits (approximately 45 minutes to 1 hour in length). A forced titration dosing strategy will be used starting with 18 mg/day OROS-MPH for 3 days, increasing to 36mg/day for the next three days; increasing to 54 mg/day in week two, and to 72 mg/day in week three through the remainder of the study (as tolerated). Participants will also attend weekly CBT sessions (approximately 1 hour in length) targeting their drug use.
- Methylphenidate (Placebo): Methylphenidate (OROS-MPH) - Placebo : Participants will be scheduled for weekly medication and research assessment visits (approximately 45 minutes to 1 hour in length). A forced titration dosing strategy will be used starting with 18 mg/day OROS-MPH placebo for 3 days, increasing to 36mg/day for the next three days; increasing to 54 mg/day in week two, and to 72 mg/day in week three through the remainder of the study (as tolerated). Participants will also attend weekly CBT sessions (approximately 1 hour in length) targeting their drug use.
Period: Overall Study
Arm/Group | Methylphenidate | Methylphenidate (Placebo)
Started | 151 | 152
Completed | 118 | 109
Not Completed | 33 | 43
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Lost to Follow-up | 9 | 17
Not completed — Moved from area | 3 | 1
Not completed — Practical Problems | 2 | 3
Not completed — Incarceration | 4 | 5
Not completed — Pressure/advice from Outsiders | 1 | 1
Not completed — Feels treatment not necessary, not worki | 0 | 1
Not completed — Other | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Methylphenidate (Placebo) | Total
Number analyzed (Participants) | 151 | 152 | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 151 | 152 | 303
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 16.4 (1.3) | 16.6 (1.2) | 16.5 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 35 | 64
  Male | 122 | 117 | 239
Region of Enrollment [Number; unit: participants]
  United States | 151 | 152 | 303

OUTCOME MEASURES:

1. Primary Outcome: ADHD Severity
Description: DSM IV ADHD Rating Scale (ADHD-RS) adolescent informant, ascertained at baseline and weekly throughout the 16 week study. This scale is an 18-item symptom checklist of self-reported adolescent ADHD symptoms. Symptoms are scored as None (0), Mild (1), Moderate (2), and Severe (3), with a summary total of scores for the 18 symptoms. Possible scores range from 0 to 54, with higher scores indicating greater severity. Outcome is measured as the decrease in total severity score over time.
Time Frame: baseline and 20 weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Methylphenidate (Placebo)
Number analyzed (Participants) | 151 | 152
units on a scale | -20.6 (11.1) | -21.8 (11.9)

2. Primary Outcome: Substance Use
Description: The change in number of days of substance use from baseline to end of the trial. The number of days of non-tobacco drug/alcohol ascertained using standard timeline follow back (TLFB) procedures.
Time Frame: 20 weeks
Population: All randomized participants.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Methylphenidate | Methylphenidate (Placebo)
Number analyzed (Participants) | 151 | 152
days | -5.7 (0.8) [-7.4 to -4.0] | -5.2 (0.9) [-7.0 to -3.5]

3. Secondary Outcome: OROS-MPH Abuse Liability
Description: Assessed by pill counts in conjunction with weekly review of subjects' medication diaries and self-reported medication compliance.
Time Frame: 20 weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | Methylphenidate | Methylphenidate (Placebo)
Number analyzed (Participants) | 151 | 152
pills | 15.4 (18.7) | 9.7 (11.2)

4. Secondary Outcome: Substance Use Outcomes
Description: The mean number of negative urine drug screens (UDS).
Time Frame: 20 weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: negative UDS
Arm/Group | Methylphenidate | Methylphenidate (Placebo)
Number analyzed (Participants) | 151 | 152
negative UDS | 3.8 (4.9) | 2.8 (4.2)

ADVERSE EVENTS:
Arm/Group | Methylphenidate | Methylphenidate (Placebo)
Serious Adverse Events (participants affected / at risk) | 4/151 | 7/152
Other Adverse Events (participants affected / at risk) | 70/151 | 64/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate (N=151) | Methylphenidate (Placebo) (N=152)
Aggression (Psychiatric disorders) | 1 (1) | 2 (2)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Cyst Rupture (General disorders) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate (N=151) | Methylphenidate (Placebo) (N=152)
Headache (Nervous system disorders) | 70 (141) | 64 (116)
Nasopharyngitis (Infections and infestations) | 23 (31) | 23 (27)
Viral Infection (Infections and infestations) | 18 (27) | 14 (24)
Upper Respiratory Tract Infection (Infections and infestations) | 12 (13) | 13 (14)
Influenza (Infections and infestations) | 5 (6) | 11 (14)
Contusion (Injury, poisoning and procedural complications) | 20 (25) | 12 (14)
Excoriation (Injury, poisoning and procedural complications) | 14 (14) | 4 (6)
Skin Laceration (Injury, poisoning and procedural complications) | 5 (6) | 12 (12)
Joint Sprain (Injury, poisoning and procedural complications) | 7 (8) | 9 (10)
Abdominal Pain Upper (Gastrointestinal disorders) | 25 (35) | 26 (35)
Vomiting (Gastrointestinal disorders) | 16 (18) | 14 (16)
Toothache (Gastrointestinal disorders) | 10 (11) | 10 (10)
Nausea (Gastrointestinal disorders) | 8 (8) | 9 (9)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 21 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 19 (22)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 15 (18)
Insomnia (Psychiatric disorders) | 21 (33) | 18 (21)
Aggression (Psychiatric disorders) | 6 (7) | 12 (16)
Nervousness (Psychiatric disorders) | 12 (15) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 12 (16) | 15 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 9 (10)
Fatigue (General disorders) | 4 (4) | 11 (11)
Decreased Appetite (Metabolism and nutrition disorders) | 25 (33) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No